CLINICAL TRIAL: NCT04744974
Title: A Randomized Clinical Trial to Assess the Impact of a Remotely Administered Diet Intervention on Symptom Burden and Inflammatory Cytokines in Myeloproliferative Neoplasm: Feasibility Phase
Brief Title: Remotely Administered Diet Intervention to Impact Symptom Burden in Myeloproliferative Neoplasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Angela G. Fleischman, Associate Professor, Division of Hematology/Oncology, Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-5932; 20-49 (Other: Chao Family Comprehensive Cancer Center)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Mediterranean or Dietary Approaches to Stop Hypertension (DASH) diet
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet (Experimental): Participants will be given dietician counseling on a Mediterranean diet
  Interventions: Behavioral: Diet intervention
- DASH diet (Experimental): Participants will be given dietician counseling on a DASH diet
  Interventions: Behavioral: Diet intervention

INTERVENTIONS:
Behavioral: Diet intervention — Participants will be given dietician counseling on their assigned diet

SUMMARY:
Myeloproliferative Neoplasm (MPN) is a chronic blood cancer without cure. The major clinical issues in MPN are 1) an increased risk of blood clots 2) symptoms thought to be driven by chronic inflammation which in some cases can be debilitating and 3) progression to acute leukemia. The current management of MPN focuses on preventing blood clots and relieving symptoms. However, treatments that reduce symptoms such as JAK inhibitors are limited to late stage MPN patients and have significant side effects including immunosuppression, reduction in platelets, and increased risk of skin cancer. Therefore, low risk interventions are sorely needed for MPN patients that can reduce symptoms. Diet represents a low risk way to reduce inflammation, specifically a Mediterranean diet has been found to reduce inflammation in cardiovascular disease. There has been a recently completed clinical trial that demonstrated MPN patients can adopt a Mediterranean diet if given dietician counseling and curriculum. However, in order to reach a larger group of people a fully remotely administered study is necessary. This is a feasibility study to determine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 with a diagnosis of a Philadelphia chromosome negative Myeloproliferative Neoplasm (MPN) including Essential Thrombocythemia (ET), Polycythemia Vera (PV), or Myelofibrosis (MF)
* Has access to the internet and email
* MPN-Total Symptom Score (MPN-TSS) score of ≥10 on screening survey
* Mediterranean Adherence score of ≤10 on screening survey
* English fluency (intervention requires conversations with study staff)
* In the opinion of the study team is amenable to changing one's diet

Exclusion Criteria:

* Pregnant or planning to become pregnant over the course of the study
* Has food allergies, intolerances, or other dietary restrictions which would severely limit changes to their diet toward a Mediterranean style diet (such as allergies to ALL tree nuts or olive oil)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
MPN Symptom Assessment form (MPN-SAF) | 16 weeks
  validated survey tool to assess symptom burden in MPN

CONTACTS AND LOCATIONS:
Overall Officials: Angela G. Fleischman, MD PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States